CLINICAL TRIAL: NCT04882943
Title: COllaboration REsearch on Chronic Cough (COREC): a French Multicenter Database
Acronym: COREC
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0378; 2020-A02774-35 (Other: ID-RCB)
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with unexplained or refractory chronic cough: Patients with cough lasting for more than 8 weeks (duration corresponding to the definition of chronic cough)
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Quality of life questionnaires

SUMMARY:
Chronic cough (TC), defined by a duration exceeding 8 weeks, is a particularly frequent symptom with a prevalence observed at 9.6% 1. Chronic cough is the cause of a major handicap for patients with a impact on their quality of life 2.

Although CT is common, management is often delicate and complex. In studies, asthma, gastroesophageal reflux disease, posterior flushing, rhino-sinusitis, or taking tussigenic medications are common causes of chronic coughs. However, chronic refractory or unexplained cough, which corresponds to cough for which no cause has been found or the treatments directed against the cause of the cough have not made it possible to resolve the cough, is a real problem in practice. nick3.

There is currently no prospective data in France on the characteristics of chronic cough (etiologies, response to treatment) and the percentage of refractory cough.

The aim of the study is to constitute a French prospective multicenter hospital cohort of chronic cough patients in order to identify, for the first time in France in a prospective and multicenter manner, the frequency of patients with refractory cough among chronic cough patients.

DETAILED DESCRIPTION:
Visit V1: Visit as part of the treatment After obtaining no objection, the patient will complete cough questionnaires

Visit V2: Visit as part of the treatment Visit carried out at 3 months with evaluation of the cough on the criteria of severity and quality of life. An evaluation of the response to treatments initiated at visit V1 will be carried out.

Visit V3: Visit as part of the treatment Visit carried out at 6 months either by telephone if response to treatment at 3 months (at the discretion of the investigators) or in the investigative center if no response to treatment at 3 months. An evaluation of the cough on the criteria of severity and quality of life will be performed.

Visit V4 to V8: Visit within the framework of research Phone call every 6 months made by a research technician. Patient severity and quality of life questionnaires will be issued in advance and completed at the time of telephone contact.

The end of research visit corresponds to the V8 visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Consultation motivated by cough lasting for more than 8 weeks (duration corresponding to the definition of chronic cough)
* Patient covered by a National Health Insurance

Exclusion Criteria:

* Active smoker or recent smoking cessation (within the past 6 months)
* Intake of medications causing cough (the patient can be included 4 weeks after treatment discontinuation if cough persists)
* Pregnant or breast-feeding women
* Upper or lower respiratory tract infection within the past 4 weeks
* Active lung disease (such as interstitial lung disease, lung cancer, abnormal dilation of the bronchi).
* History of chronic bronchitis.
* Current treatment with an angiotensin converting enzyme (ACE) inhibitor
* History of cancer within the past 5 years or active cancer (excluding cutaneous squamous-cell carcinoma).
* Person not fluent in French
* Adult not able to express his/her consent verbally
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic cough patients
Sampling Method: Non-Probability Sample
Enrollment: 576 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
French prospective multicenter hospital cohort of chronic cough patients (requency of patients with unexplained or refractory chronic cough (URCC) | 24 months
  set up a French prospective multicenter hospital cohort of chronic cough patients in order to identify the frequency of patients with unexplained or refractory chronic cough (URCC) for the first time in France

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GUILLEMINAULT, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No